CLINICAL TRIAL: NCT00198757
Title: Efficacy of 2 Diet Plans Designed for People With Type II Diabetes on Weight and Health Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Medifast, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDI2002-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-05

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

INTERVENTIONS:
Behavioral: Medifast Plus for Diabetics Meal Replacement Supplements
Behavioral: Standard ADA recommended diet for type 2 diabetics

SUMMARY:
The objective of this study is to evaluate the efficacy of Medifast Plus for Diabetics compared to a standard weight loss treatment program, in terms of changes in weight loss in overweight men and women over an 86 week active weight loss and weight maintenance program. There will be up to 34 weeks active weight loss and 52 weeks weight maintenance. The planned sample size is 80 overweight (BMI 25-40) males and females aged 18-65 with type 2 diabetes. It is anticipated that pre-packaged meal replacements will provide an advantage to those desiring weight loss.

DETAILED DESCRIPTION:
This study will test the efficacy of Medifast Plus for Diabetics compared to a standard American Diabetes Association (ADA) weight loss treatment program using whole foods in 80 participants (randomized into 2 groups of 40) during an active weight loss and weight maintenance program lasting 68-86 weeks. The study data collection will occur in two phases, active weight loss (phase 1) and weight maintenance (phase 2). Transition into phase 2 will be individually timed by participant attainment of a goal 'healthy' weight following a minimum of 16 weeks, or week 34, whichever comes first. A dietitian will prescribe an individualized weight loss and weight maintenance calorie levels for participants based on the Harris Benedict equation (RMR x AF x Deficit; RMR=resting metabolic rate, AF=activity factor). All participants will have a goal 'healthy' weight determined at baseline by a combination of personal participant goals, Harris Benedict equation predictions, body composition goals, and BMI range, but in no case will participants be prescribed a goal weight that would result in an BMI of less than 24. For the weight loss phase, participants will be randomly assigned to one of 2 groups, Medifast Plus for Diabetics or standard ADA weight loss treatment program. Both groups will attend educational lessons every other week during weight loss, and once every four weeks during the maintenance phase. Data collection visits will occur when goal weight is reached, at week 26 of maintenance, and week 52 of maintenance. During the weight loss phase, group 1 will receive 5 Medifast Plus for Diabetics supplements and one small meal to consume every day. As participants reach their goal weights, they will be re-randomize according to weight loss success and gender categories into two different maintenance plans. One maintenance group will first receive 26 weeks of Medifast Plus for Diabetics maintenance diet, still receiving 5 supplements/day but with a larger portion of calories coming from whole foods, followed by 26 weeks of a purely food-based maintenance diet (the same as the control group, where participants will choose all foods and receive no supplements). The second group will be a reversal of the order of maintenance diets (first the food-based maintenance for 26 weeks, and then the Medifast Plus for Diabetics maintenance for 26 weeks). The control group will remain on a food-based, no supplement maintenance diet for the entire 52-week maintenance period. Participants will be encouraged to report any adverse events or changes in medications at any time during the study

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years of age.
2. Overweight (Body Mass Index between 25-40) and desiring weight loss
3. Normal ECG (electrocardiogram) or abnormalities deemed medically acceptable (no acute ischemic changes or V-tach, eg)
4. Not using appetite-affecting medications (e.g., Prozac or other SSRIs, synthroid, steroids) unless on established and stable dose
5. Not using weight loss drugs (phentermine, sibutramine, orlistat, eg)
6. Willing and able to comply with the protocol requirements
7. Willing and able to give informed consent
8. Have a regular source of health care and permission of primary care provider
9. Using an acceptable method of birth control (tubal ligation, abstinence, properly used condom or diaphragm, oral or implanted contraceptives, or intrauterine device) for women of childbearing potential

Exclusion Criteria:

1. Chronic uncontrolled health problems (not including obesity and diabetes). Participants may not have bulimia, laxative abuse, substance abuse, alcohol intake > 10 drinks per week, or have an uncontrolled psychiatric disorder (major depression, bipolar disorder, etc), as determined at screening
2. Breast-feeding or pregnant at screening by serum pregnancy test if female of childbearing capacity. To be considered not childbearing potential, participant must be at least one year post-menopausal or surgically sterile

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-07; Study Completion 2005-01

PRIMARY OUTCOMES:
Body weight (change from baseline through attaining goal or week 34,
at 26 weeks of maintenance,
at 52 weeks of maintenance

SECONDARY OUTCOMES:
percent body fat (at baseline vs. at attainment of goal weight or at week 34, and at weeks 26 and 52 of maintenance,
blood pressure,
blood values including hemoglobin A1C, glucose, cholesterol, and triglycerides;
changes in medication costs and health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health